CLINICAL TRIAL: NCT07231731
Title: Association of MicroRNA-151-5p Expression With Systemic Inflammatory Response and Cognitive Status in Patients After Coronary Artery Bypass Surgery (MiRNACOG)
Brief Title: Dynamics of microRNA Expression and Systemic Inflammatory Response in POCD After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Visnja Ikic, MD, Doctor of medicine, Specialist in anaesthesiology, reanimatology and intensive care medicine, Subspecialist in intensive care medicine, Osijek University Hospital
Other Study IDs: microRNA-POCD
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Biomarkers; Coronary Artery Bypass Surgery; Interleukin-6; MicroRNAs; Postoperative Cognitive Complications; Systemic Inflammatory Response Syndrome
Keywords: Anesthesia, General; Blood-Brain Barrier; Cardiac Surgical Procedures; Cardiopulmonary Bypass; Cholinesterases; Cognitive Disorders; Cognitive Dysfunction; Coronary Artery Bypass; Coronary Artery Disease; Critical Care; Extracorporeal Circulation; Gene Expression; Inflammation; Interleukins; Mental Disorders; Myocardial Revascularization; Nervous System Diseases; Neurocognitive Disorders; Neuroinflammatory Diseases; Neuropsychological Tests; Pathological Conditions, Signs and Symptoms; Pathologic Processes; Perioperative Period; Postoperative Care; Postoperative Cognitive Complications; Postoperative Complications; S100B protein, human; Thoracic Surgery; Treatment Outcome
MeSH Terms: conditions — Postoperative Cognitive Complications; Systemic Inflammatory Response Syndrome; Cognitive Dysfunction; Coronary Artery Disease; Inflammation; Mental Disorders; Nervous System Diseases; Neurocognitive Disorders; Neuroinflammatory Diseases; Pathological Conditions, Signs and Symptoms; Pathologic Processes; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — MicroRNA expression will be determined from serum isolated from a venous blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Bypass Graft (CABG) group: The study include a cohort of patients, between the ages of 65 and 80, who undergo coronary artery bypass graft surgery to treat coronary artery disease, receiving 2 or more coronary artery bypass grafts with the use of extracorporeal circulation.

SUMMARY:
Postoperative cognitive decline (POCD) is one of the most common complications after cardiac surgery. It is characterized by impaired memory, attention, and executive functions and can have long-term consequences. The goal of this observational study was to investigate the mechanisms of cognitive decline after cardiac surgery and potential biomarkers that could aid in the diagnosis, prevention, and treatment of POCD. The investigators focused on the role of microRNAs (miRNAs) and systemic inflammatory response to surgery, extracorporeal circulation, and anesthesia as potential factors involved in the development of the neuroinflammatory response and subsequent POCD. The main question this study aims to answer is whether perioperative miRNA 151-5p expression is associated with POCD after surgery. The second aim is to examine the association between miRNA-151-5p and systemic inflammation. The investigators measured circulating miRNA-151-5p levels and plasma levels of inflammatory biomarkers in patients undergoing surgical myocardial revascularization. To assess cognitive function, participants completed the Montreal Cognitive Assessment (MoCA Test). Changes in the measured values of miRNA-151-5p expression and inflammatory markers, as well as changes in cognitive status after surgery, were assessed in relation to the preoperative state.

DETAILED DESCRIPTION:
Surgical myocardial revascularization is a procedure used in patients with ischemic heart disease to bypass atherosclerotic narrowings or blockages of the coronary arteries using an arterial or venous graft (Coronary Artery Bypass Grafting - CABG). One of the most common complications after cardiac surgery is postoperative cognitive decline (POCD). It is characterized by impaired memory, attention, and executive functions and can have long-term consequences, such as delayed physical therapy and mobilization, prolonged stay in the intensive care unit and hospital, more frequent discharge to nursing homes, reduced quality of life, and increased mortality.

The causes of POCD are multifactorial. The systemic inflammatory response to surgery, extracorporeal circulation, and anesthesia is considered a factor in the development of the neuroinflammatory response and subsequent POCD. Neuroinflammation can cause dysfunction or death of brain cells and damage to the blood-brain barrier, leading to an increase in the level of biochemical markers of brain injury in the blood. Studies indicate that numerous microRNAs (miRNAs) play a role in controlling the inflammatory response. MiRNAs are small, endogenous, non-coding RNA molecules, typically 18-25 nucleotides long, that regulate gene expression at the post-transcriptional level. They are central mediators of cellular proliferation, differentiation, and apoptosis. MiRNA levels in tissues and peripheral blood are similar, and circulating miRNAs are stable and suitable for measurement. Specific miRNAs (miRNA 151-5p, 505, 499, 625, and others) may be potential early biomarkers of brain damage after a mild traumatic brain injury. Anesthesia and surgery also, through complex mechanisms, can cause changes in brain cells that can lead to the release of specific miRNAs, and these miRNAs can be detected in blood and various biological fluids.

Hypothesis: Higher levels of perioperative miRNA-151-5p expression are associated with the systemic inflammatory response and with the development of POCD.

Aim of this study is:

1. To investigate the association between miRNA-151-5p expression levels and biochemical parameters of systemic inflammation, as well as the association of both with cognitive status in patient undergoing CABG surgery.
2. To investigate the association between patients' demographic and clinical characteristics and miRNA-151-5p expression levels, the level of biochemical parameters of systemic inflammation, and patients' cognitive status.

Research plan:

The research was carried out at the Clinical Hospital Centre Osijek. Respecting the inclusion and exclusion criteria for participation in the study, the research included patients aged 65 to 80 years who, according to the American Society of Anesthesiologists (ASA) classification, are classified into groups III and IV, and who are undergoing CABG surgery with the use of extracorporeal circulation. Surgeries were performed according to the standard protocol for balanced anesthesia, cardiac surgery, and extracorporeal circulation. All participants underwent the same anesthetic procedure and anesthesia based on midazolam, propofol, sufentanyl, rocuronium and sevoflurane. The depth of anesthesia was monitored using Patient State Index (PSI). All surgeries were performed using extracorporeal circulation with the maintenance of normothermia (36 °C).

Blood samples for determination of levels of cholinesterase, interleukin-6, protein S100B, miRNA-151-5p expression and routine laboratory parameters (complete blood count, levels of troponin I, C-reactive protein, procalcitonin, glucose, urea, creatinine, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, total bilirubin, albumin, electrolytes, lactate, coagulation tests, and arterial blood gas analysis) were taken at three time points: before surgery prior to induction of anesthesia, immediately after the procedure upon admission to the intensive care unit, and 48 hours after the surgical procedure.

Cognitive function testing was performed the day before surgery and postoperatively, once daily every day until the 6th postoperative day. The investigators used a validated scoring scale for assessing cognitive functions, the Montreal Cognitive Assessment - MoCA Test. Demographic and clinical data were recorded for all subjects. Subjects were followed up 7 days.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing coronary artery bypass graft surgery to treat coronary artery disease
* two or more coronary bypass surgery with the use of extracorporeal circulation
* patients between the ages of 65 and 80
* patients according to the classification of the American Society of Anesthesiologists (ASA) classified in groups III and IV
* patients who agreed to participate in the research and signed an informed consent

Exclusion Criteria:

* patients with communication difficulties (severe visual, hearing and speech impairment)
* illiterate patients
* patients with a history of dementia, schizophrenia, Parkinson's disease, Alzheimer's disease, alcoholism
* patients with previously known liver failure of any grade according to the Child-Pough classification
* patients with previously known renal failure greater than grade 2
* patients taking immunosuppressive, corticosteroid and anticholinergic therapy
* intraoperatively used cell-saver and/or hemofilter
* patients in whom the planned procedure is not performed
* patients in whom it is not possible to assess cognitive functions postoperatively (patients sedated due to intra- or postoperative surgical complications)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing coronary artery bypass grafting surgery at the Department of Cardiac and Thoracic Surgery of the Clinic for Surgery, Clinical Hospital Center Osijek.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Perioperative changes in microRNA 151-5p expression. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  MicroRNA-151-5p expression levels will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU. Levels of microRNA expression will be calculated relative to reference microRNA-16-5p using 2-∆∆cT method.
Perioperative changes in cognitive function measured by Montreal Cognitive Assessment (MoCA Test). | 1 day before surgery and once daily postoperatively, up to the 6th postoperative day.
  Cognitive function will be assessed in all patients at enrollment one day before surgery, and daily for the following six postoperative days using the Montreal Cognitive Assessment (MoCA test).
  Montreal Cognitive Assessment scale: minimum score is 0 and maximum score is 30 points, a score of 26 or above is considered normal, while scores below this may indicate cognitive impairment. A score of 18-25 suggests mild cognitive impairment, 10-17 suggests moderate impairment, and a score 0-9 suggests severe impairment.

SECONDARY OUTCOMES:
Perioperative changes in levels of white blood cells. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission.
  Levels of white blood cells will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Perioperative changes in levels of C-reactive protein. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  Levels of C-reactive protein will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Perioperative changes in levels of procalcitonin. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  Levels of procalcitonin will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Perioperative changes in levels of interleukin-6. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  Levels of interleukin-6 will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Perioperative changes in levels of cholinesterase. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  Levels of cholinesterase will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Perioperative changes in levels of protein S-100B. | Preoperative, within 2 hours of ICU admission, 48 hours after ICU admission
  Levels of protein S-100B will be measured in tree time points: preoperative before induction of anaesthesia, postoperative within 2 hours of Intensive Care Unit (ICU) admission and 48 hours after admission to the ICU.
Patient demographic data. | From enrollment to the end of cognitive testing at 6th postoperative day.
  Patient demographic data: age, gender, education, and previous medical history will be recorded and correlated with microRNA expression levels, inflammatory biomarkers and the Montreal Cognitive Assessment (MoCA test) scores.
  Montreal Cognitive Assessment scale: minimum score is 0 and maximum score is 30 points, a score of 26 or above is considered normal, while scores below this may indicate cognitive impairment. A score of 18-25 suggests mild cognitive impairment, 10-17 suggests moderate impairment, and a score 0-9 suggests severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, Professor, Study Chair — University Hospital Osijek
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
After study completion, upon reasonable request, data may be shared with other researchers.

REFERENCES:
- [Background] van Harten AE, Scheeren TW, Absalom AR. A review of postoperative cognitive dysfunction and neuroinflammation associated with cardiac surgery and anaesthesia. Anaesthesia. 2012 Mar;67(3):280-93. doi: 10.1111/j.1365-2044.2011.07008.x. PMID 22321085
- [Background] Kok WF, Koerts J, Tucha O, Scheeren TW, Absalom AR. Neuronal damage biomarkers in the identification of patients at risk of long-term postoperative cognitive dysfunction after cardiac surgery. Anaesthesia. 2017 Mar;72(3):359-369. doi: 10.1111/anae.13712. Epub 2016 Dec 17. PMID 27987229
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Greaves D, Psaltis PJ, Ross TJ, Davis D, Smith AE, Boord MS, Keage HAD. Cognitive outcomes following coronary artery bypass grafting: A systematic review and meta-analysis of 91,829 patients. Int J Cardiol. 2019 Aug 15;289:43-49. doi: 10.1016/j.ijcard.2019.04.065. Epub 2019 Apr 24. PMID 31078353
- [Background] Kapoor MC. Neurological dysfunction after cardiac surgery and cardiac intensive care admission: A narrative review part 1: The problem; nomenclature; delirium and postoperative neurocognitive disorder; and the role of cardiac surgery and anesthesia. Ann Card Anaesth. 2020 Oct-Dec;23(4):383-390. doi: 10.4103/aca.ACA_138_19. PMID 33109792
- [Background] Polito F, Fama F, Oteri R, Raffa G, Vita G, Conti A, Daniele S, Macaione V, Passalacqua M, Cardali S, Di Giorgio RM, Gioffre M, Angileri FF, Germano A, Aguennouz M. Circulating miRNAs expression as potential biomarkers of mild traumatic brain injury. Mol Biol Rep. 2020 Apr;47(4):2941-2949. doi: 10.1007/s11033-020-05386-7. Epub 2020 Mar 26. PMID 32219772
- [Background] Pozniak T, Shcharbin D, Bryszewska M. Circulating microRNAs in Medicine. Int J Mol Sci. 2022 Apr 3;23(7):3996. doi: 10.3390/ijms23073996. PMID 35409354
- See also: MoCA - Cognitive Assessment [Internet]. [cited 2022 Feb 9]. MoCA - Cognitive Assessment. Available from: https://www.mocatest.org/. — https://www.mocatest.org